CLINICAL TRIAL: NCT07360015
Title: Radiographic Evaluation of Bone Level Evaluation Around Implants in All on Four Hybrid OT Restorations With Different Number of Screws
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Egyptian Russian University (Network); Fayoum University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FD-ERU-Rec 25
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss in Jaw
Keywords: implant-supported prostheses; OT abutments; crestal bone loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 screws (Experimental): screw retained implant supported mandibular prosthesis with OT Equator abutments (3 screws).
  Interventions: Other: OT Equator abutments with 3 screws.
- 4 screws (Experimental): screw retained implant supported mandibular prosthesis with OT Equator abutments (4 screws).
  Interventions: Other: OT Equator abutments with 4 screws.

INTERVENTIONS:
Other: OT Equator abutments with 3 screws. — screw retained implant supported mandibular prosthesis with OT Equator abutments (3 screws).
  Arms: 3 screws
Other: OT Equator abutments with 4 screws. — screw retained implant supported mandibular prosthesis with OT Equator abutments (4 screws).
  Arms: 4 screws

SUMMARY:
This research aims to compare between using OT Equator abutments for constructing implant supported fixed mandibular prosthesis with different number of screws (3 screws vs 4 screws) regarding the marginal bone height alteration around the implants through radiographic evaluation.

DETAILED DESCRIPTION:
Fourteen completely edentulous male patients free from any systemic diseases that would affect bone metabolism, had no history of recent administration of chemotherapy or radiotherapy and no history of para-functional habits will be selected from out-patients clinic.

The first group will include seven patients who will be planned to receive screw retained implant supported mandibular prosthesis with OT Equator abutments (3 screws).

The second group will include seven patients who will be planned to receive screw retained implant supported mandibular prosthesis with OT Equator abutments (4 screws).

Pre-surgical protocol:

For each patient, upper and lower complete dentures will be constructed. Using dual CBCT scan protocol, stereolithographic surgical guide will be constructed according to virtual implant planning in the software, and the 3D surgical guide will be used to insert four implants in mandibular canines and mandibular first molar positions.

OT EQUATOR abutments will be screwed to the four implants. Denture conversion was done for temporization:

After three months of implant insertion, the final prosthesis will be constructed and then screwed to the OT Equator abutments.

For the first group one screw will be avoided and the final prosthesis will be screwed to the OT Equator abutments with 3 screws only.

For the second group and the final prosthesis will be screwed to the OT Equator abutments with 4 screws.

The DIGORA Optime intraoral sensor and a specially built acrylic template for each patient will be used to take intraoral radiographs with the standardized long cone paralleling technique to measure changes of crestal bone level around each implant. Periods of 0 (immediately after delivery of final prosthesis), 3, 6, and 9 months after delivery of final prosthesis for radiographic evaluation. Bone loss measurements will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients
* male patients
* free from any systemic diseases
* no history of recent administration of chemotherapy or radiotherapy
* no history of para-functional habits

Exclusion Criteria:

* female patients
* diabetic patients and patients with bone metabolism diseases
* history of recent administration of chemotherapy or radiotherapy
* history of para-functional habits
* Heavy smokers.
* Heavy consumption of Alcohol

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients were only selected to avoid the effect of sex related variations as habits and physiology. Also, to avoid the effect of sex related hormonal changes which were reported to contribute to mucosal changes and osteoporosis.
Enrollment: 14 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
crestal bone loss around implants | 12 months
  The DIGORA Optime intraoral sensor and a specially built acrylic template for each patient will be used to take intraoral radiographs with the standardized long cone paralleling technique to measure changes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine - Egyptian Russian University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided